CLINICAL TRIAL: NCT02176252
Title: A Phase I, Double-blind, Placebo Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects in Healthy Male and Female Japanese Subjects After Single and Multiple Doses (Bid) of AZD1722
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamic of AZD1722 in Healthy Male and Female Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5611C00005
Record Dates: First submitted 2013-11-11; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD1722 (Experimental): Dose escalation from 5 mg to 90 mg BID
  Interventions: Drug: AZD1722; Drug: Placebo

INTERVENTIONS:
Drug: AZD1722
  Other Names: RDX5791; Tenapanor
Drug: Placebo

SUMMARY:
The study is designed to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of AZD1722 in healthy Japanese subjects at increasing doses given for 7 days in order to allow for including Japanese subjects in future global studies. A cohort of Caucasian subjects will be included in the study to evaluate cardiac effects, assessed by digital ECGs (dECG) recordings, also in Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman
* Body mass index between 18 and 29.9 kg/m2, inclusive

Exclusion Criteria:

* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the gastrointestinal (GI) tract
* Any surgery on the small intestine or colon, excluding appendectomy
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, metabolic, endocrine, neurologic, psychiatric disease, or any condition that may interfere with the subject successfully completing the trial or that would present a safety risk to the subject.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 3 weeks
  Measurement of safety laboratories, ECGs, vital signs, and physical exams

SECONDARY OUTCOMES:
pharmacodynamic activity | up to one week
  24-hour stool sodium and phosphorus
pharmacokinetics | up to one week
  plasma drug concentration to calculate AUC, if possible

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Director — Ardelyx, Inc.
Locations (1):
- WCCT Global, Cypress, California, United States

REFERENCES:
- [Derived] Johansson S, Rosenbaum DP, Knutsson M, Leonsson-Zachrisson M. A phase 1 study of the safety, tolerability, pharmacodynamics, and pharmacokinetics of tenapanor in healthy Japanese volunteers. Clin Exp Nephrol. 2017 Jun;21(3):407-416. doi: 10.1007/s10157-016-1302-8. Epub 2016 Jul 1. PMID 27368672